CLINICAL TRIAL: NCT02959320
Title: A Randomized Clinical Trial of Direct Anterior vs. Anterolateral Approach for Hip Arthroplasty After Femoral Neck Fracture in the Senior Population
Brief Title: Direct Anterior vs. Anterolateral Approach for Hip Arthroplasty After Femoral Neck Fracture in the Senior Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William W. Cross, III M.D., Assistant Professor of Orthopedics,, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-003695
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Anterior Approach (Active Comparator): All patients receiving a hip hemiarthroplasty through a Direct Anterior Approach (DAA) will have their surgeries performed with the aid of fluoroscopy on an OSI Hana table that allows the operative limb to be manipulated through range of motion and traction while keeping the pelvis stabilized. This table also has a radiolucent platform about the pelvis, enabling the surgery to be fluoroscopically assisted. The incision for the DAA will extend from a proximal point about 2 cm distal and 2 cm lateral to the ASIS to a point 8-12 cm distal and slightly lateral to this.
  Interventions: Procedure: Hip Hemiarthroplasty
- Anterolateral Approach (Active Comparator): All patients receiving a hip hemiarthroplasty through an the Anterolateral Approach (ALA) will have their surgeries performed on a standard OR table in a contralateral lateral decubitus position. With the leg in the position of sleep, a straight 8-12 cm incision will be made, centered over the greater trochanter and femoral shaft with 1/3 of the incision extending superior to the tip of the greater trochanter.
  Interventions: Procedure: Hip Hemiarthroplasty

INTERVENTIONS:
Procedure: Hip Hemiarthroplasty — This single-institution, prospective, randomized clinical trial will be performed on consecutive elderly patients admitted for surgical treatment of displaced femoral neck fractures with hemiarthroplasty (HA).

SUMMARY:
Displaced femoral neck fractures are one group of hip fracture patients that are commonly treated with cemented hemiarthroplasty (HA) or total hip arthroplasty (THA). In the elective hip arthroplasty population, the direct anterior approach (DAA) has shown to be effective in helping patients to quickly obtain high postoperative function. This approach has also been shown to be effective in arthroplasty for displaced femoral neck fractures in a few studies. However, the only studies that directly compare two approaches for hip arthroplasty for femoral neck fractures utilize the anterolateral approach (ALA) versus posterior approach (PA) or DAA versus PA. No studies of which we are aware directly compare the DAA to the ALA. The DAA and ALA are the two most popular approaches for bipolar hemiarthroplasty at our institution, so we are setting out to determine the differences between them.

DETAILED DESCRIPTION:
Displaced femoral neck fractures are one group of hip fracture patients that are commonly treated with cemented hemiarthroplasty (HA) or total hip arthroplasty (THA). Compared to those who receive a THA, recipients of HA tend to be less active, more debilitated, and more dependent on gait aids and the care of others. In this population, the increased stability and decreased operating time associated with HA is thought to be more important than the minimal increase in function this population could achieve with THA. Additionally, cemented femoral stems in HA are thought to result in less pain, increased function, and less periprosthetic fracture risk when compared to cementless stems.

With the relative pre-injury debility of the femoral neck fracture population, especially those receiving HA, it is important to optimize all aspects of patient care to allow them to participate in therapy and return them to their preoperative functional level as quickly as possible. Furthermore, any intervention in this population should minimize the physiologic insult of surgery as much as possible. In the elective hip arthroplasty population, the direct anterior approach (DAA) has shown to be effective in helping patients to quickly obtain high postoperative function. This approach has also been shown to be effective in arthroplasty for displaced femoral neck fractures in a few studies. However, the only studies that directly compare two approaches for hip arthroplasty for femoral neck fractures utilize the anterolateral approach (ALA) versus posterior approach (PA) or DAA versus PA. No studies of which we are aware directly compare the DAA to the ALA. The DAA and ALA are the two most popular approaches for bipolar hemiarthroplasty at our institution, so investigators are setting out to determine the differences between them.

ELIGIBILITY:
Inclusion Criteria:

* isolated displaced femoral neck fracture (AO type 31-B2 and 31 B3)
* age≥65 years
* preinjury ambulation with or without a gait aid
* surgical intervention ≤ 48 hours after fracture.

Exclusion Criteria:

* age <65 years
* patients with other fractures or dislocations
* wheelchair bound
* >48 hours between fracture and surgery, presence or history of infection, active metastatic disease, previous ipsilateral hip prosthesis
* active major psychiatric illness
* active drug or alcohol abuse
* BMI >40, and actively failing contralateral hip prosthesis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-11; Primary Completion 2021-09-07 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Number of patients showing improvement using the Timed Up and Go (TUG) Test | Baseline to 12 months
  Purpose of test is to assess mobility and will be administered by a nurse who is blinded to the surgical approach.

CONTACTS AND LOCATIONS:
Overall Officials: Cross W. William, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials